CLINICAL TRIAL: NCT05673005
Title: MED3000 Topical Gel for On-Demand Treatment of Post-Radical Prostatectomy Erectile Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Martin Kathrins, M.D., Assistant Professor of Surgery, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021P002976
Record Dates: First submitted 2021-12-08; First posted 2023-01-05 (Actual); Results first posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-11

CONDITIONS: Erectile Dysfunction Following Radical Prostatectomy

STUDY DESIGN:
Intervention Model Description: Medical device (MED3000)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- MED3000 topical gel treatment (Experimental): All qualified enrolled patients will receive treatment with MED3000 topical gel on demand through the 12-week follow-up visits.
  Interventions: Device: MED3000 topical gel

INTERVENTIONS:
Device: MED3000 topical gel — Topical gel that has been shown to improve erectile dysfunction when used as needed.

SUMMARY:
The investigators are doing this research to evaluate the efficacy and safety of topical MED3000 therapy in men with persistent erectile dysfunction 1.5 to 4 years following radical prostatectomy surgery.

DETAILED DESCRIPTION:
MED3000 is a topical gel that has been developed to treat patients with erectile dysfunction. The investigators postulate that on demand treatment with MED3000 can improve on-demand erectile function among men status-post radical prostatectomy, allowing for some endogenous cavernosal nerve function recovery for 1.5 to 4 years post-surgery among men with normal baseline pre-surgical erectile function.

ELIGIBILITY:
Inclusion Criteria:

* Men who underwent robotic bilateral nerve-sparing radical prostatectomy between 18 and 36 months prior to study commencement
* Subjects are 18-48 months status-post radical prostatectomy
* Subjects have any degree of erectile dysfunction based on IIEF questionnaire
* Age 40 - 70 at study commencement
* Diagnosed with low/intermediate-risk prostate cancer:

  * PSA < 20 ng/ml
  * Gleason score =< 8
  * Prostate Cancer stage =< T3a
* Normal pre-radical prostatectomy erectile function (IIEF >=26) or equivalent response on EPIC
* Baseline erectile dysfunction at time of screening (despite use of erectogenic aids of any kind) and enrolment following washout (IIEF-ED domain <=25)
* Sexually active, in a stable heterosexual relationship for at least 6 months prior to screening
* Able to understand and complete patient questionnaires
* Serum prostate specific antigen (PSA) undetectable (no evidence of disease recurrence)
* Able to consent to participate
* Documented written informed consent from both patient and his female partner

Exclusion Criteria:

* Anatomical abnormalities in the genitalia or pelvic region such as severe phimosis
* Post-Radical Prostatectomy complications that could impact safety or effectiveness of medical therapy for erectile function (treatment for pelvic hematoma, urinary or intestinal fistula, unresolved anastomotic leak)
* Tumor upstaging beyond T3a
* Incomplete / sub-total nerve sparing on either side
* Previous or scheduled treatment with pelvic salvage radiotherapy and/or androgen deprivation therapy
* Prior receipt of androgen deprivation therapy
* Any other condition that would prevent the patient from completing the study, as judged by the Principal Investigator

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kathrins, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 patients met all the eligibility criteria and enrolled in the study.
Period: Overall Study
Arm/Group | MED3000 Topical Gel Treatment
Started | 20
Completed | 17
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: 1 patient did not meet enrollment criteria
Arm/Group | MED3000 Topical Gel Treatment
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (4.6)
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 1 patient did not meet inclusion criteria
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 2
    White | 18
    More than one race | 0
    Unknown or Not Reported | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: one subject did not meet enrollment criteria
  Participants
    Female | 0
    Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Whether the Erectile Function Domain of the International Index of Erectile Function Mean Change From Baseline Met or Exceeded the Minimally Clinically Important Difference (MCID) of 4
Description: To investigate the effect of MED3000 topical gel for treatment of erectile dysfunction after nerve sparing prostatectomy (based on Erectile Function domain of the International Index of Erectile Function) (units on a scale) and whether it met MCID criteria of change of mean 4 [IIEF EF minimum score is 0, maximum score is 75, with higher scores representing improved erectile function); units on a scale
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: IIEF-EF difference (units on scale)
Arm/Group | MED3000 topical gel treatment
Number analyzed (Participants) | 17
IIEF-EF difference (units on scale) | 0.8 (3.9) [1 to 11]

2. Secondary Outcome: Efficacy of MED3000 Topical Gel (Self-Esteem and Relationship Questionnaire)
Description: The efficacy of MED3000 in patients at weeks 4, 8 and 12 using:
  The change from baseline in Self-Esteem and Relationship (SEAR) questionnaire for men (units on a scale) [SEAR minimum score is 0, maximum score is 70, with higher scores representing improved outcomes); units on a scale
Time Frame: 12 weeks
Reporting Status: Not Posted

3. Secondary Outcome: The Change From Baseline in Urinary Incontinence Using the Expanded Prostate Cancer Index Composite (EPIC) (Efficacy)
Description: The efficacy of MED3000 in patients at weeks 4, 8 and 12 (units on a scale) [EPIC minimum score 18; maximum score 93, with higher scores representing improved function]
Time Frame: 12 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Change From Baseline in All Domains of the IIEF.
Description: The efficacy of MED3000 in patients at weeks 4, 8 and 12 (units on a scale)
Time Frame: 12 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Efficacy of MED3000 Topical Gel on Post-prostatectomy Incontinence
Description: The change from baseline in 24 hour pad weight and usage number per day at 12 weeks. (grams)
Time Frame: 12 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Efficacy of MED3000 Topical Gel on Stretched Flaccid Penile Length
Description: The change from baseline of the stretched flaccid penile length following 12-weeks of treatment
Time Frame: 12 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Adverse Events of MED3000 Topical Gel
Description: Treatment-related adverse events in male patients and female partners occurring during treatment with MED3000.
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up
Description: No adverse events, local reactions, or difficulty with application reported by any participant over the 12-week period.
Arm/Group | MED3000 Topical Gel Treatment
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/05/NCT05673005/Prot_SAP_000.pdf